CLINICAL TRIAL: NCT06744803
Title: The Effect of a Gamified Neuropathy Management Application on Cancer Behavior in Cancer Patients Undergoing Chemotherapy: A Prospective Follow-Up Study
Brief Title: The Effect of a Gamified Neuropathy Management Application on Cancer Behavior in Cancer Patients Undergoing Chemotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Betül Çakmak, PhD, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01.08.2024/78 KARAR NO:36
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Chemotherapy Induced Pain Neuropathy; Nursing; Gamification
Keywords: cancer; chemotherapy induced pain neuropathy; nursing; gamification
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized control trial (prospective follow up study)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Gamified Neuropathy Management Application
  Interventions: Behavioral: Gamified Neuropathy Management Application on Cancer Behavior
- control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Gamified Neuropathy Management Application on Cancer Behavior — The study will be conducted in three phases:
  Phase 1: The content of the gamified neuropathy management application used in the study will be prepared by the researchers using relevant literature.
  Phase 2: The developed gamified neuropathy management application will be introduced to patients during one-on-one interviews at the daytime chemotherapy clinic. After collecting pre-test data, the application will be sent to the patients, who will be asked to use it for 8 weeks.
  Phase 3: Following the start of the study's implementation, patients will be contacted in the 4th and 8th weeks to collect mid-study and post-test data.
  Other Names: intervention group
  Arms: intervention group

SUMMARY:
This study will be conducted to determine the effect of a gamified neuropathy management application on cancer behavior in cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Cancer patients may experience treatment-related issues throughout their treatment process. Chemotherapy-induced peripheral neuropathy is one of the symptoms that negatively affects patients' overall health status. Peripheral neuropathy can occur during or after chemotherapy, leading to sensory, motor, and autonomic nerve damage. It is particularly common among cancer patients receiving taxane- and platinum-based chemotherapy.

Effective management of neuropathy is a crucial aspect of nursing care. Here are some key points regarding this issue: pharmacological and non-pharmacological methods, lifestyle control, and nursing interventions are employed. The management of peripheral neuropathy can have a significant impact on the overall health and well-being of cancer patients undergoing chemotherapy. Nurses play a vital role in this process by providing support that enhances patients' quality of life and improves treatment outcomes.

Gamification applications, which have recently started to be used in patient education, represent a contemporary approach. However, no studies have been found utilizing gamification specifically in patient education for cancer. For this reason, this study aims to contribute to patients' neuropathy management using a gamification application.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing chemotherapy treatment and have completed their first cycle.
* Literate (able to read and write).
* Able to use a smartphone.
* Aged between 18 and 65 years.
* Willing to participate in the study voluntarily.

Exclusion Criteria:

* Participants who do not use the application during the study period
* Participants who fail to complete the data collection forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of gamified neuropathy management application on chemotherapy-associated peripheral neuropathic pain. | 6 months
  DN4 Questionnaire: The DN4 pain questionnaire, developed by the French neuropathic pain group, is a questionnaire that includes symptoms and findings associated with neuropathic pain. The individual being evaluated answers the questions with yes or no. The total scale score is calculated by giving 1 point for each yes answer and 0 point for each no answer. In the scale, the cutoff value for neuropathic pain is determined as 4/10 and above. Turkish validity and reliability was determined by Unal-Çevik et al. It was made by and the Cronbach alpha coefficient was 0.97; The specificity and sensitivity in diagnosing neuropathic pain were found to be 96.6% and 95%, respectively.
The effect of gamified neuropathy management application on chemotherapy-associated peripheral neuropathic level | 6 months
  CIPNAT, Tofthagen et al. (2011b). CIPNAT, which is a Likert type scale, consists of 2 parts. The first part consists of 36 items asking about symptom frequency, severity, and discomfort. In the second part, there are 14 items that evaluate which of the daily living activities peripheral neuropathy affects. First, patients are asked whether any of the nine symptoms developed after chemotherapy treatment. The frequency, severity and discomfort of the symptoms experienced after each question answered "Yes" are scored and evaluated with a 0-10 numerical rating scale. If the answer to the first 4 questions on the scale is "No", the other questions are not continued. These questions are the questions that determine whether there is the presence of CBPN (Kutlutürkan et al. 2017). A high score from the scale indicates that CBPN is high. The Turkish validity and reliability study of the scale was conducted by Kutlutürkan et al. (2017). The Cronbach alpha coefficient of the scale is 0.970.
The effect of gamified neuropathy management application on cancer behaviour | 6 months
  Heitzmann et al. Developed by KSI-KV in 2011. This inventory is a 12-item unidimensional measurement tool designed to assess cancer patients' self-efficacy in coping. Each item of this 12-item scale is scored between 1-9. The scale score is calculated as the sum of all items. High scores from the scale indicate high self-efficacy for coping. The Cronbach alpha coefficient of this scale, which was evaluated on three sample groups, was found to be a = 0.84, a = 0.84, a = 0.88 for each sample, respectively. The construct validity of the scale was conducted using Exploratory Factor Analysis for the first sample, and four factors were obtained according to the results of the analysis: (1) Maintaining Independence and Positive Attitude; (2) Participating in Medical Care; (3) Coping and Stress Management; (4) Managing Affect. Adaptation of this scale to Turkish was made by İyigün et al. (2017).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I have not discussed this with other researchers